CLINICAL TRIAL: NCT05521711
Title: TRADE Trial - Tree Nut Immunotherapy Route Development and Evaluation
Acronym: TRADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: AAAAI Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HAH-21-013
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Tree Nut Allergy; Food Allergy
Keywords: Immunotherapy; Randomized Controlled Trial (RCT)
MeSH Terms: conditions — Nut Hypersensitivity; Food Hypersensitivity | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active low dose oral immunotherapy and Placebo sublingual immunotherapy (Experimental)
  Interventions: Other: Food
- Placebo low dose oral immunotherapy and Active sublingual immunotherapy (Experimental)
  Interventions: Other: Food
- Placebo low dose oral immunotherapy and Placebo sublingual immunotherapy (Experimental)
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Commercially available powders or liquids

SUMMARY:
Tree nut immunotherapy Route Assessment and DEvelopment (TRADE) is a randomized controlled trial that evaluates the efficacy and safety of sublingual immunotherapy and lower, more tolerable, doses of oral immunotherapy than currently in use.

ELIGIBILITY:
Inclusion Criteria:

* Allergic to tree nut with baseline threshold of 444 mg protein or less and provides consent, and where applicable, assent.

Exclusion Criteria:

1. History of anaphylaxis to tree nut severe enough to cause shock, syncope, or intubation
2. Eosinophilic or other inflammatory gastrointestinal disease within the past 2 years
3. Severe (GINA severity class 5) or uncontrolled asthma including exacerbation within past 6 months
4. Use of biologics, other food immunotherapy or experimental treatment in past 6 months.
5. Ongoing other allergic diseases severe enough to preclude discontinuing antihistamines for 7 days prior to assessment visits
6. Pregnancy or significant medical condition (e.g., liver, kidney, gastrointestinal, cardiovascular, hematologic, or pulmonary disease; allergy to the oat-based placebo) which would put the participant at excessive risk for food allergic reactions as judged by local investigator

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Eliciting dose thresholds to food challenge | 1 year

SECONDARY OUTCOMES:
Quality of life | 1 Year
  Food allergy quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Derek Chu, MD PhD FRCPC, Principal Investigator — Hamilton Health Sciences & McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Will consider on a case by case basis.